CLINICAL TRIAL: NCT03805776
Title: Role of Intermittent Fasting in Improving High Density Lipoprotein Cholesterol
Brief Title: Intermittent Fasting in Dyslipidemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, NASEER AHMED, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 123
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Intermittent Fasting; Dyslipidemias; HDL Cholesterol, Low Serum; Hepatic Enzymes and Function Abnormalities; Anemia; Kidney Diseases; Cardiac Function
Keywords: Intermittent fasting; Fasting; Cholesterol
MeSH Terms: conditions — Intermittent Fasting; Dyslipidemias; Hypoalphalipoproteinemias; Anemia; Kidney Diseases; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Will observe intermittent fasting
  Interventions: Other: Fasting (diet restruction for specific period)
- Control (No Intervention)

INTERVENTIONS:
Other: Fasting (diet restruction for specific period) — 12-14 hours fasting
  Arms: Interventional

SUMMARY:
World Health Organization report notifies of the escalating global burden of cardiovascular diseases (CVD), projecting that it will become the major worldwide cause of death and disability by 2020. The South Asian countries have the highest rates of CVD globally. It is widely acknowledged that South Asians have 40-60% higher risk of CVD linked to mortality, compared with other populations. Multiple human population studies have established the concentration of high density lipoprotein (HDL) cholesterol as an independent, inverse predictor of the risk of having a cardiovascular event. Furthermore, HDLs have several well-documented functions with the potential to protect against cardiovascular disease. This study trial is designed to find out the role of intermittent fasting to improve the dyslipidemia and particularly increase the levels of HDL in general population. Investigators expect that the intermittent fasting will significantly enhance the level of HDL and reduce cardiovascular events in general population.

DETAILED DESCRIPTION:
INTRODUCTION:

Overall lipid profile is important in cardiovascular diseases but particularly serum HDL levels have long been recognized as an independent inverse prognostic marker of CVD, when the Framigham study, in 1980s showed that HDL below 40-60mg/dl is of prognostic relevance. A rise of 1mg/dl in HDL levels is considered to reduce coronary artery disease (CAD) risk to 2-3%. Even patients with elevated total cholesterol (TC) and LDL, presenting a high HDL are seen to be protected from atherosclerosis. Multiple human population studies have shown the concentration of HDL cholesterol as an independent, inverse predictor of the risk of having a cardiovascular event. Additionally, HDL has several well-documented functions with the potential to protect against cardiovascular diseases. These include an ability to promote the efflux of cholesterol from macrophages in the artery wall, inhibit the oxidative modification of LDL, inhibit vascular inflammation, inhibit thrombosis, promote endothelial repair, promote angiogenesis, anti-oxidant, enhance endothelial function, improve diabetic control, and inhibit hematopoietic stem cell proliferation. HDL also exerts direct cardio protective effect, which are mediated with its interactions with the myocardium.

Various studies have emphasised the high incidence of CVD within the South Asian countries. The increased risk of cardiovascular events in South Asians at a younger age might be due to unknown factors affecting plaque rupture, the interaction between prothrombotic factors and atherosclerosis, or may be due to any undiscovered risk factors. Urbanisation and westernisation is characterised by a distinct increase in the intake of energy dense foods, a decrease in physical activity, and a heightened level of psychosocial stress, all of which promote the development of hyperglycaemia, hypertension, and dyslipidaemia. Most common dyslipidaemia in South Asians is low HDL-C and high triglycerides. High triglyceride and low HDL-C levels are metabolically interlinked. This metabolic phenotype is also associated with increased levels of small LDL particles despite relatively normal levels of LDL-C among South Asians. This clinical syndrome is accompanied by insulin resistance, a condition frequently referred to as atherogenic dyslipidemia, which is a common metabolic derangement among Asian. South Asians not only have lower HDL levels but also have a higher concentration of small, less-protective HDL particles. One proposed mechanism is presence of dysfunctional HDL particles. Another potential explanation for the apparent blunted cardioprotection of HDL in South Asians might be related to HDL particle size. Small particles might be less efficient in reverse cholesterol transport. In general, HDL particle size tends to be lower in patients with CHD and those with low HDL-C levels . Alarmingly, an estimated 60-80% of Pakistani population has been reported to have low HDL. There are a number of non-pharmacological and pharmacological recommendations for management of low HDL. Non-pharmacological (functional food) strategies are reported to increase HDL levels around 10-15% and which include regular exercise , body weight reduction in obese individuals , cessation of cigarette smoking in smokers and dietary modifications like decrease intake of saturated trans-fatty acids with increase intake of omega-3 polyunsaturated fatty acids . There are also a number of pharmacological agents being considered as therapeutic options but the tolerability and safety issues limit their use in addition to limited success in improving HDL. IF may be a dietary method to aid in the improvement of the lipid profile in healthy, obese and dyslipidemia men and women, reducing total cholesterol, LDL, triglycerides and increasing HDL levels. However, the majority of studies that analyze the IF impacts on the lipid profile and body weight loss are observational and lack detailed information about diet. Randomized clinical trials with larger sample size are needed to evaluate the IF effects mainly in population with dyslipidemia.

HYPOTHESIS:

Intermittent fasting is capable of improving dyslipidemia and particularly enhancement of serum, HDL which can increase the cardioprotection in high risk general population.

OBJECTIVES:

To evaluate the effect of intermittent fasting on cholesterol levels specifically on HDL.

DATA STORAGE AND MANAGEMENT:

Every participant will be given a code number, all data will be saved according to the code numbers. Privacy will be maintain of each and every participant. Records will be kept confidential and used only for scientific purposes by authorized personnel. The hard copies will be kept in locked cupboards and soft data will be managed in password protected computers. Data will be stored at institutional level for almost 15 years.

DISSEMINATION OF FINDINGS AND PUBLICATION PLAN:

Investigators expect that Ajwa and intermittent fasting will significantly improve HDL levels in order to enhance the cardiac protection. This research will help in promoting the significance of use of functional food and fasting to improve overall health. Investigators expect at least two publications from this study. The findings of the study will be presented in international conference and will be published in well reputed journal.

ELIGIBILITY:
Inclusion Criteria:

* General population with serum HDL less than 40 mg/dl for men and women
* Adult ages 18- 80 years will be included in the study.

Exclusion Criteria:

* Individuals Patients already observing fasting regularly
* Pregnant women and individuals with diabetes, metabolic syndrome or any other co-morbidity will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
Lipid profile | 6 weeks
  Change in HDL more than 3mg/dl Change in LDL more than 3mg/dl Cholesterol and TG
weight loss | 6 weeks
  Change in body weight (kg), as measured by scale weight
Blood pressure | 6 weeks
  Reduction in systolic and diastolic

SECONDARY OUTCOMES:
Fasting Glucose | 6 weeks
  Fasting glucose mg/dl
Fasting Insulin | 6 weeks
  Fasting insulin (IU/L)
Waist circumference Waist circumference (cm) | 6 weeks
  WC in cm
Lipid profile HbA1c (%) Lipids | 6 weeks
  Total cholesterol (mg/dl), LDL cholesterol (mg/dl), HDL cholesterol (mg/dl), and triglycerides (mg/dl)
Waist circumference | 6 weeks
  Waist circumference (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Aksungar FB, Eren A, Ure S, Teskin O, Ates G: Effects of intermittent fasting on serum lipid levels, coagulation status and plasma homocysteine levels. Annals of nutrition & metabolism 2005, 49:77-82. 2. Ahmet I, Wan R, Mattson MP, Lakatta EG, Talan M: Cardioprotection by intermittent fasting in rats. Circulation 2005, 112:3115-3121. 3. Santos HO, Macedo RCO: Impact of intermittent fasting on the lipid profile: Assessment associated with diet and weight loss. Clinical nutrition ESPEN 2018, 24:14-21. 4. Adlouni A, Ghalim N, Saı̈le R, Hda N, Parra H-J, Benslimane A: Beneficial effect on serum apo AI, apo B and Lp AI levels of Ramadan fasting. Clinica Chimica Acta 1998, 271:179-189. 5. Hammouda O, Chtourou H, Aloui A, Chahed H, Kallel C, Miled A, Chamari K, Chaouachi A, Souissi N: Concomitant effects of Ramadan fasting and time-of-day on apolipoprotein AI, B, Lp-a and homocysteine responses during aerobic exercise in Tunisian soccer players. PloS one 2013, 8:e79873.
- [Derived] Ahmed N, Farooq J, Siddiqi HS, Meo SA, Kulsoom B, Laghari AH, Jamshed H, Pasha F. Impact of Intermittent Fasting on Lipid Profile-A Quasi-Randomized Clinical Trial. Front Nutr. 2021 Feb 1;7:596787. doi: 10.3389/fnut.2020.596787. eCollection 2020. PMID 33598473